CLINICAL TRIAL: NCT06195956
Title: Effects of Lower Limb Kinetic Chain Exercise to Shoulder Rehabilitation Program in Patients With Shoulder Impingement Syndrome
Brief Title: The Effect of Lower Limb Kinetic Chain Exercise in Shoulder Impingement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, the effect of lower limb kinetic chain exercise in shoulder impingement, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: kinetic chain exercise
Record Dates: First submitted 2023-12-25; First posted 2024-01-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder Impingement Rehabilitation (Active Comparator): rehabilitation program consisting of strengthening exercises (for scapular stabilizers and rotator cuff) and stretching exercises (for pectoralis major, pectoralis minor, latissimus dorsi, levator scapula).
  Exercises done 3 times per weeks, 3 repetitions per exercise for 3 months
  Interventions: Other: exercise
- Shoulder Impingement Rehabilitation with LL KC Exercise (Experimental): rehabilitation program consisting of strengthening exercises (for scapular stabilizers and rotator cuff) and stretching exercises (for pectoralis major, pectoralis minor, latissimus dorsi, levator scapula) in addition to lower limb kinetic chain exercise.
  Exercises done 3 times per weeks, 3 repetitions per exercise for 3 months
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Exercises done 3 times per weeks, 3 repetitions per exercise for 3 months

SUMMARY:
The goal of this clinical trial study is to investigate the effect of performing lower limb kinetic chain exercise on muscle activation of scapular muscle strength ratio in patients with shoulder impingement. the main question it aims to answer is:

Does the addition of lower limb kinetic chain exercise to a shoulder exercise program improve scapular muscles strength ratio in patients with shoulder impingement? participants will be devided into two groups to be compared: The first group will be given a rehabilitation program consisting of strengthening exercises (for scapular stabilizers and rotator cuff) and stretching exercises (for pectoralis major, pectoralis minor, latissimus dorsi, levator scapula) The second group will be given the same exercises in addition to lower limb kinetic chain exercise

DETAILED DESCRIPTION:
The term "kinetic chain" (KC) describes the sequential activation of body segments during functional movement patterns (Wilk et al., 2016). An effective KC will produce, summate, and enable effective mechanical energy transmission along the entire chain, which will support function. Any link in the KC that is inefficient has the potential to adversely affect force transfer to nearby segments (Ben kibler et al., 2000 & Martic et al., 2014). Consequently, therapists usually recommend incorporating trunk and lower extremity movements into shoulder rehabilitation programs in order to maximize efficient energy transfer throughout the entire KC (Sciascia et al., 2012 & Magarey et al., 2003). Thus, the investigators hypothesize that adding a lower limb (LL) kinetic chain exercise to a shoulder exercise program will improve scapular muscles strength ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges between 20 and 45 years old
* Unilateral shoulder pain lasting more than 6 weeks
* At least one positive finding in each of these categories:

  1. Painful arc of movement during flexion or abduction
  2. Positive Neer or Hawkins-Kennedy impingement signs
  3. Pain on resisted lateral rotation, abduction or Jobe test

Exclusion Criteria:

* History of surgery
* History of fracture or dislocation
* Type III acromion
* Rotator cuff tear
* Long head of biceps tendon tear
* Cervical radiculopathy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography to evaluate the activation patterns, timing and ratio of scapular muscles during movement | baseline
  EMG activity of the three trapezius parts (upper, middle and lower) and Serratus anterior will be evaluated.
  1. Electrodes for registration of upper trapezius activity are placed halfway between the spinous process of C7 and the posterior acromion.
  2. Electrodes for registration of middle trapezius activity are placed halfway on the horizontal line between the thoracic spine and the root of the scapular spine.
  3. Electrodes for registration of Lower trapezius activity are placed obliquely upward and laterally along a line between the intersection of the scapular spine with the vertebral border of the scapula and the seventh thoracic spinous process.
  4. Electrodes for registration of Serratus Anterior activity are applied anterior to the latissimus dorsi and posterior to the pectoralis major

SECONDARY OUTCOMES:
Shoulder pain and disability Index | baseline
  To test pain and functional disability before and after interventions. 0-20: mild shoulder pain and disability 21-40: moderate shoulder pain and disability 41-60: severe shoulder pain and disability 61-80: very severe shoulder pain and disability 81-100: extremely severe shoulder pain and disability

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Melhat, Phd, Study Director — Cairo University
Locations (1):
- Outpatient physical therapy, Faculty of physical therapy, Giza, Egypt

REFERENCES:
- [Background] Wilk KE, Arrigo CA, Hooks TR, Andrews JR. Rehabilitation of the Overhead Throwing Athlete: There Is More to It Than Just External Rotation/Internal Rotation Strengthening. PM R. 2016 Mar;8(3 Suppl):S78-90. doi: 10.1016/j.pmrj.2015.12.005. PMID 26972270
- [Background] Sciascia A, Thigpen C, Namdari S, Baldwin K. Kinetic chain abnormalities in the athletic shoulder. Sports Med Arthrosc Rev. 2012 Mar;20(1):16-21. doi: 10.1097/JSA.0b013e31823a021f. PMID 22311288